CLINICAL TRIAL: NCT04512638
Title: A Multicenter Randomized Controlled Open-label Trial of Conservative Management Versus Minimally Invasive Treatment With Leukocyte- and Platelet-rich Fibrin Versus Primary Surgery in Patients With Newly Diagnosed Osteonecrosis of the Jaw
Brief Title: Best Treatment Choice for Osteonecrosis of the Jaw
Acronym: BETCON
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tim Van den Wyngaert (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor-Investigator, Tim Van den Wyngaert, Principal Investigator, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/11482/1; 338 (Registry Identifier: EDGE)
Record Dates: First submitted 2020-08-08; First posted 2020-08-13 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Medication Related Osteonecrosis of the Jaw
MeSH Terms: interventions — Anti-Bacterial Agents; Amoxicillin; Chlorhexidine; Minimally Invasive Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conservative treatment (Active Comparator): Amoxicillin-based antibiotics and chlorhexidine oral rinse. Minor debridement. Primary wound closure is not part of this treatment strategy.
  Interventions: Drug: Antibiotics; Drug: Chlorhexidine mouthwash
- Minimally invasive approach + LPRF (Experimental): Amoxicillin-based antibiotics and chlorhexidine oral rinse. Minimally-invasive surgical treatment, including sequestrectomy, debridement of soft tissue, and application of LPRF membranes before tension-free wound closure is obtained. Marginal resection of all necrotic bone is not part of this treatment strategy.
  Interventions: Drug: Antibiotics; Drug: Chlorhexidine mouthwash; Procedure: Minimally invasive surgery with LPRF
- Primary surgical management (Experimental): Amoxicillin-based antibiotics and chlorhexidine oral rinse. Removal of the necrotic bone without excessive resection of healthy bone. Buccal mucoperiosteal flaps will be used to achieve a tension-free mucosal coverage.
  Interventions: Drug: Antibiotics; Drug: Chlorhexidine mouthwash; Procedure: Surgical resection

INTERVENTIONS:
Drug: Antibiotics — Antibiotic treatment is the same in all groups.
  Monotherapy for 4 weeks with:
  No penicillin contra-indication
  * Amoxicillin-clavulanate 875mg tid PO Penicillin contra-indication or intolerance
  * Clindamycin 300mg tid PO
  After 4 weeks patients will be switched to consolidation antibiotics:
  No penicillin contra-indication
  * Amoxicillin 1g bid PO Penicillin contra-indication or intolerance
  * Clindamycin 300mg tid PO
  Antibiotic treatment can be discontinued after 4 weeks when the MRONJ lesions has healed.
  Other Names: amoxicillin
Drug: Chlorhexidine mouthwash — Patients in all treatment groups will be prescribed aqueous chlorhexidine 0.12% tid rinse for 2 weeks, with subsequent switch to 0.05% for the duration of the study or until healing of the MRONJ lesion has occurred.
  Other Names: chlorhexidine
Procedure: Minimally invasive surgery with LPRF — Minimally-invasive surgical treatment, including sequestrectomy, debridement of soft tissue, and application of LPRF membranes before tension-free wound closure is obtained. Marginal resection of all necrotic bone is not part of this treatment strategy.
  Arms: Minimally invasive approach + LPRF
Procedure: Surgical resection — Primary surgical management consisting of the removal of the necrotic bone without excessive resection of healthy bone. Buccal mucoperiosteal flaps will be used to achieve a tension-free mucosal coverage.
  Arms: Primary surgical management

SUMMARY:
BETCON is a pragmatic randomized controlled open-label multi-center study in patients with newly diagnosed stage I-II MRONJ designed to answer the question whether minimally invasive management with LPRF membranes or primary surgical treatment is better than the standard of care of conservative therapy alone. The primary end-point is the time to mucosal healing. Secondary end-points consist of supporting measures of efficacy, patient reported symptoms, quality of life, well-being, and functioning.

DETAILED DESCRIPTION:
While effective for symptom control and well tolerated, conservative treatment of MRONJ yields highly variable mucosal healing rates ranging between 20 to 50%. In an effort to improve these suboptimal outcomes, many adjunct treatment modalities have been studied, of which the use of minimally invasive surgery with autologous platelet rich plasma (LPRF) to improve wound healing has attracted considerable attention, with reported mucosal closure rates of up to 86% in single arm case series. More recently, improved understanding of the need for pre-operative infection control and adaptation of surgical protocols has renewed the interest in the primary surgical treatment of MRONJ with mucosal closure achieved in up to 90% of patients in some case series.

Therapeutic studies of MRONJ have almost exclusively focused on mucosal healing as the desired end-point of MRONJ treatment, with little or no attention to patient symptoms, quality of life, functioning and well-being during treatment, even though the resolution of MRONJ symptoms and limiting treatment related adverse events may be equally important to patients.

This comparative effectiveness research (CER) study is a randomized controlled open-label multi-center study in patients with newly diagnosed stage I-II MRONJ and is designed to answer the question whether minimally invasive treatment with LPRF membranes or primary surgical treatment improves outcomes when added to the standard of care of conservative treatment alone. The study also incorporates pragmatic design elements and uses patient reported outcomes (PRO) to determine which treatment offers the best humanistic outcomes considering both efficacy and measures of quality of life, functioning, well-being and symptom control. Indeed, this study will not use an investigational new drug (or drug regimen), device, or surgical technique, but rather evaluate their relative efficacy to guide future clinical management. Finally, plasma and saliva will be collected to identify prognostic and predictive biomarkers of outcome.

ELIGIBILITY:
Inclusion criteria:

* >18 years of age
* Provision of signed informed consent
* A history of at least one administration of, or an ongoing treatment with, a bone modifying agent in dose registered for the prevention of skeletal related events in bone metastatic disease or multiple myeloma
* Diagnosis of stage I-II MRONJ according to AAOMS 2014 criteria not more than 8 weeks prior to the date of screening

Exclusion criteria:

* Any prior treatment for MRONJ other than local antiseptic rinses, systemic antibiotics, or analgesics
* Prior radiotherapy to the head and neck region
* Medical contraindication to receive any of the possible study treatments
* Stage III MRONJ characterized by very extensive bone necrosis, pathological fracture, or fistulas to the skin or sinuses
* Multiple MRONJ lesions that cannot be closed in a single surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Time to confirmed mucosal healing | 12 months
  Time after randomization until the observation of healed mucosa (without presence of surgical suturing material) at the site of MRONJ, with a first observation of healed mucosa requiring confirmation after 4 weeks.

SECONDARY OUTCOMES:
Mucosal closure | 6 months
  Proportion of patients with mucosal closure 6 months after randomization
Time to MRONJ healing | 12 months
  Time to resolution of MRONJ symptoms after start of treatment
Relapse rate of MRONJ | 12 months
  Incidence of patients with relapse at the site of MRONJ
Antibiotics use | 12 months
  Total duration of exposure to antimicrobial agents
Evolution of cancer health-related quality-of-life | 12 months
  Changes over time as measured with the EORTC QLQ-C30 questionnaire.
Evolution of general health status | 12 months
  Changes over time as measured with the EUROQOL 5D (EQ-5D-5L) questionnaire.
Evolution of oral health-specific quality-of-life | 12 months
  Changes over time as measured with the Oral Health Impacts Profile (OHIP-14) and the SWOG0702 Oral Health and Oral Health-related Quality of Life questionnaires.

OTHER OUTCOMES:
Treatment related adverse events | Through study completion, an average of 1 year
  Incidence and intensity of treatment emergent adverse events
Quality-adjusted Time Without Symptoms and Toxicity (Q-TWiST) | Through study completion, an average of 1 year
  This analysis analysis considers three health states: toxicity, time without symptoms and toxicity (TWiST), and relapse. The toxicity state comprises the total time after randomization and before relapse of MRONJ symptoms spent with toxicity, regardless of when the toxicity started or gaps between toxicities. The TWiST state is defined as the time of relapse of MRONJ symptoms minus time with toxicities. The duration of the relapse state is defined as overall survival time minus time to relapse of MRONJ symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Van den Wyngaert, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (4):
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
  - AZ Nikolaas, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beth-Tasdogan NH, Mayer B, Hussein H, Zolk O, Peter JU. Interventions for managing medication-related osteonecrosis of the jaw. Cochrane Database Syst Rev. 2022 Jul 12;7(7):CD012432. doi: 10.1002/14651858.CD012432.pub3. PMID 35866376
- See also: Trial website — http://www.betcon.be